CLINICAL TRIAL: NCT05366907
Title: Open Cholecystectomy Among Patients Undergoing Laparoscopic Cholecystectomy in a Tertiary Care Centre: A Descriptive Cross-Sectional Study
Brief Title: Open Cholecystectomy Among Patients Undergoing Laparoscopic Cholecystectomy.
Status: Completed | Type: Observational
Sponsor: Chitwan Medical College (Other)
Responsible Party: Principal Investigator, Gaurav Katwal, Principal Investigator, Chitwan Medical College
Other Study IDs: CMC-IRC/0770798-271
Record Dates: First submitted 2022-05-03; First posted 2022-05-09 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cholelithiasis; Laparoscopic Cholecystectomy; Cholecystectomy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is done — It is a descriptive cross-sectional study so no groups like case/controls are present. All the cases are included in the study.

SUMMARY:
In the current era, laparoscopic cholecystectomy is the treatment of choice for symptomatic gallstone disease. The aim of this study is to find out the prevalence of open cholecystectomy among patients undergoing laparoscopic cholecystectomy in a tertiary care center.

DETAILED DESCRIPTION:
Laparoscopic Cholecystectomy (LC) is the gold standard surgery for symptomatic cholelithiasis with low mortality and morbidity.1,2 However, 1% to 15% of conversion rate to Open Cholecystectomy (OC) during laparoscopic cholecystectomy has been reported.3 Converted cases were associated with increased perioperative time, complication rates, perioperative costs, the length of hospital stay, and a higher 30-day readmission rate.3,4 Conversion was also associated with complications including bile leak, bile duct injury, or bleeding, requiring reoperation or transfusion, and death. A recent detailed critical review found that preoperative variables like male gender, older age, high body mass index, previous abdominal surgery, the severity of cholecystitis, and gallbladder wall thickness were associated with the higher rate of conversion to OC.4 However, data regarding its prevalence lacking in our setting.

The aim of this study is to find out the prevalence of open cholecystectomy among patients undergoing laparoscopic cholecystectomy in a tertiary care centre.

ELIGIBILITY:
Inclusion Criteria:

* All the cases of Symptomatic Cholelithiasis elected for Laparoscopic Cholecystectomy

Exclusion Criteria:

* Age <10 years,
* Gall Bladder Malignancy,
* Adults with preoperative choledocholithiasis, and
* Perforated gall bladder

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the cases of elective LC admitted at the Department of Surgery at CMCTH were included.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Laparoscopic to Open cholecystectomy | 1 year
  Demographic details, previous attack of biliary pathology, underlying condition, Huang classification of the biliary system are collected. And conversion rate among these patients were calculated with CR= number of converted surgeries/(number of converted surgeries + number of LC surgeries) × 100) Objectives- To identify the prevalence of conversion rate and, To compare the CR among independent variables- Age, Sex, history of previous attack with dependent variable Open cholecystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Harish Chandra Neupane, MS, Study Chair — CMCTH
Locations (1):
- Chitwan Medical College Teaching Hospital, Bharatpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
Data can be provided to the individual interested researcher only on the basis of sound interest in research with good moral intention.

REFERENCES:
- [Background] Genc V, Sulaimanov M, Cipe G, Basceken SI, Erverdi N, Gurel M, Aras N, Hazinedaroglu SM. What necessitates the conversion to open cholecystectomy? A retrospective analysis of 5164 consecutive laparoscopic operations. Clinics (Sao Paulo). 2011;66(3):417-20. doi: 10.1590/s1807-59322011000300009. PMID 21552665
- [Background] Aziret M, Karaman K, Ercan M, Vargol E, Toka B, Arslan Y, Oter V, Bostanci EB, Parlak E. Early laparoscopic cholecystectomy is associated with less risk of complications after the removal of common bile duct stones by endoscopic retrograde cholangiopancreatography. Turk J Gastroenterol. 2019 Apr;30(4):336-344. doi: 10.5152/tjg.2018.18272. PMID 30945646
- [Background] European Association for the Study of the Liver (EASL). Electronic address: easloffice@easloffice.eu. EASL Clinical Practice Guidelines on the prevention, diagnosis and treatment of gallstones. J Hepatol. 2016 Jul;65(1):146-181. doi: 10.1016/j.jhep.2016.03.005. Epub 2016 Apr 13. No abstract available. PMID 27085810
- [Background] Deka P, Islam M, Jindal D, Kumar N, Arora A, Negi SS. Analysis of biliary anatomy according to different classification systems. Indian J Gastroenterol. 2014 Jan;33(1):23-30. doi: 10.1007/s12664-013-0371-9. Epub 2013 Sep 5. PMID 24006122
- [Background] Shea JA, Berlin JA, Escarce JJ, Clarke JR, Kinosian BP, Cabana MD, Tsai WW, Horangic N, Malet PF, Schwartz JS, et al. Revised estimates of diagnostic test sensitivity and specificity in suspected biliary tract disease. Arch Intern Med. 1994 Nov 28;154(22):2573-81. PMID 7979854
- [Background] Coffin SJ, Wrenn SM, Callas PW, Abu-Jaish W. Three decades later: investigating the rate of and risks for conversion from laparoscopic to open cholecystectomy. Surg Endosc. 2018 Feb;32(2):923-929. doi: 10.1007/s00464-017-5767-7. Epub 2017 Aug 4. PMID 28779254
- [Background] Hu ASY, Menon R, Gunnarsson R, de Costa A. Risk factors for conversion of laparoscopic cholecystectomy to open surgery - A systematic literature review of 30 studies. Am J Surg. 2017 Nov;214(5):920-930. doi: 10.1016/j.amjsurg.2017.07.029. Epub 2017 Jul 21. PMID 28739121
- [Background] Philip Rothman J, Burcharth J, Pommergaard HC, Viereck S, Rosenberg J. Preoperative Risk Factors for Conversion of Laparoscopic Cholecystectomy to Open Surgery - A Systematic Review and Meta-Analysis of Observational Studies. Dig Surg. 2016;33(5):414-23. doi: 10.1159/000445505. Epub 2016 May 5. PMID 27160289
- [Background] van de Graaf FW, Zaimi I, Stassen LPS, Lange JF. Safe laparoscopic cholecystectomy: A systematic review of bile duct injury prevention. Int J Surg. 2018 Dec;60:164-172. doi: 10.1016/j.ijsu.2018.11.006. Epub 2018 Nov 12. PMID 30439536
- See also: DOI — https://www.nepjol.info/index.php/nmcj/article/view/30038